CLINICAL TRIAL: NCT06316960
Title: A Prospective, Multicenter Clinical Study on The Safety and Efficacy of Avapritinib in The Treatment of Relapsed/Refractory Pediatric Core Binding Factor Acute Myeloid Leukemia (CBF-AML) With KIT Mutation
Brief Title: Safety and Efficacy of Avapritinib in Relapsed or Refractory Pediatric CBF-AML With KIT Mutation
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospital of Soochow University (Other)
Responsible Party: Principal Investigator, Shaoyan Hu, Study Chair, Children's Hospital of Soochow University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AVACBFKIT
Record Dates: First submitted 2024-03-12; First posted 2024-03-19 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: AML, Childhood; Relapse/Recurrence; Refractory AML; Core Binding Factor Acute Myeloid Leukemia; C-KIT Mutation
Keywords: Avapritinib; KIT; CBF AML; Childhood; Relapsed/Refractory
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Recurrence | interventions — avapritinib; Azacitidine; Decitabine; Idarubicin; Cytarabine; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Relapsed/Refractory CBF-AML with KIT mutation (Experimental): The relapsed/refractory patients will receive a combination treatment of decitabine/azacitidine+ IdAG (idarubicine + cytarabine + granulocyte stimulating factor)regimen along with avapritinib. CBF-AML with KIT mutated patients with molecular relapse after hematopoietic stem cell transplantation may receive avapritinib combined with demethylating agents or interferon or donor lymphocyte infusion without low-dose chemotherapy. The dose of avapritinib will start at 50mg/m2/d, and if platelets stabilize at 50 ×10^9/L and neutrophils stabilize above 1.0 ×10^9/L after one week, the dose can be increased to 100mg/m2/d, with a maximum daily dose of 100mg. Avapritinib should be discontinued in the presence of febrile neutropenia or active infection, and avapritinib can be resumed once the infection is controlled, with each treatment cycle not exceeding 28 days.
  Interventions: Drug: Avapritinib; Drug: Azacitidine Injection; Drug: Decitabine Injection; Drug: Idarubicin Hydrochloride; Drug: Cytarabine; Drug: Granulocyte Colony-Stimulating Factor

INTERVENTIONS:
Drug: Avapritinib — 50mg/m2/day for weighing bodyweight >10kg, 1.65mg/kg/day for weighing ≤ 10kg, po, qd, d1-28.
  Other Names: AYVAKIT
Drug: Azacitidine Injection — 75mg/m2/d for weighing >10kg, 2.5mg/kg/d for weighing ≤ 10kg, d1-7, ivgtt, qd, more than 3 hours. Azacitidine and decitabine cannot be used simultaneously.
  Other Names: Azacitidine
Drug: Decitabine Injection — 20mg/m2/d for weighing >10kg, 0.67mg/kg/d for weighing ≤ 10kg, d1-5, ivgtt, qd, more than 3 hours. Azacitidine and decitabine cannot be used simultaneously.
  Other Names: Decitabine
Drug: Idarubicin Hydrochloride — 5mg/m2/day for weighing >10kg, 0.17mg/kg/day for weighing ≤ 10kg, d 6, 8, 10 (d 8, 10, 12 for azacitidine) ivgtt, qod, more than 1 hour at 10 am.
  Other Names: Idarubicine
Drug: Cytarabine — 10mg/m2/day for weighing >10kg, 0.33mg/kg/day for weighing ≤ 10kg, d6-15 （d8-17 for azacitidine ）, s.c., q12h.
  Other Names: CYTOSAR
Drug: Granulocyte Colony-Stimulating Factor — 300ug/day for weighing >10kg, 10ug/kg/day for weighing ≤10kg, d0-5, s.c., qd.
  Other Names: Recombinant Human Granulocyte Colony-Stimulating Factor Injection

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of avapritinib in relapsed or refractory pediatric core binding factor acute myeloid leukemia with KIT mutation.

DETAILED DESCRIPTION:
This is a multicenter, single-arm, prospective, and intervention trial. About 30% of core binding factor acute myeloid leukemia (CBF-AML) patients still relapse under current treatment. Some studies have found that KIT mutations, especially the D816V mutation, may predict relapse and decrease overall survival (OS) in CBF-AML. Avapritinib has been approved for the treatment of gastrointestinal stromal tumors with KIT or PDGFRA mutations. Avapritinib was also effective for the treatment of minimal residual disease in acute myeloid leukemia with t (8;21) and KIT mutation failing to immunotherapy after allogeneic hematopoietic stem cell transplantation in a single-center, retrospective report. 11 centers from China carry out the AVACBFKIT regimen including Avapritinib, hypomethylating agents and low dose chemotherapy for the treatment of relapsed or refractory pediatric CBF-AML with KIT mutation. The main focus of this study is to evaluate the efficacy and safety of avapritinib in the regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Gender unlimited;
2. Under 18 years;
3. Diagnosis of acute myeloid leukemia (according to the 2022 WHO classification).
4. Presence of t(8;21)/RUNX1::RUNX1T1 or inv(16)/t(16;16)/CBFβ::MYH11;
5. KIT mutation;
6. Refractory AML: AML patients who do not achieve CR or CRi after induction therapy;
7. Relapsed AML: patients who achieved remission after consolidation therapy or transplantation, FISH confirmed that the fusion gene turned positive, or extramedullary leukemia infiltration;
8. No active infections;
9. Liver function: Tbil ≤2×ULN, ALT/AST ≤3×ULN, creatinine clearance ≥50ml/min;
10. ECOG score <2;
11. Expected survival time >12 weeks;
12. Participants must have the ability to understand and be willing to participate in this study and must sign an informed consent form.

Exclusion Criteria:

1. Have received prior treatment with avapritinib;
2. Receiving other targeted therapies for AML at the same time, such as dasatinib, sorafenib, gilteritinib, venetoclax, etc;
3. Presence of active uncontrolled infection (including bacterial, fungal, or viral infection);
4. Present of significant underlying organ diseases: such as myocardial infarction, chronic heart failure, decompensated liver or kidney dysfunction；
5. With other malignancies requiring treatment；
6. Already enrolled in another interventional clinical study；
7. The researchers determined that the individual is not suitable to participate in this trial.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Composite remission rate (CRc) | The evaluation time point is day28-day35 from the start of regimen.
  Composite remission rate (CRc), including the sum of the number of patients with complete remission (CR), complete remission with partial hematologic recovery (CRh), complete remission with incomplete blood count recovery (CRi), and morphologically leukemia-free (MLFS) as a percentage of the total number of patients who participated in the efficacy analysis.

SECONDARY OUTCOMES:
Overall survival | From date of enrollment until the date of the occurrence of death or last follow-up, assessed up to 60 months.
  Overall survival (OS) was deﬁned as the date from enrollment to the date of death or last follow-up for surviving patients.
Progression-free survival | From date of enrollment until the date of disease progression, conﬁrmed relapse, or death, whichever occurred ﬁrst, assessed up to 60 months.
  Progression-free survival (PFS) was deﬁned as the date from enrollment to the date of disease progression, conﬁrmed relapse, or death, whichever occurred ﬁrst.

CONTACTS AND LOCATIONS:
Overall Officials: Shaoyan Hu, MD, PhD, Principal Investigator — Children 's Hospital of Soochow University
Locations (12):
- China (12):
  - First Affiliated Hospital Of University of Science and Technology of China, Hefei, Anhui
  - The Second Hospital of Anhui Medical University, Hefei, Anhui
  - Guangzhou Women and Children Medical Center, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - Kaifeng Children's Hospital, Kaifeng, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Third Xiangya Hospital of Central South University, Changsha, Hunan
  - XiangYa Hospital Central South University, Changsha, Hunan
  - Children's Hospital of Soochow University, Suzhou, Jiangsu
  - Xuzhou Children's Hospital, Xuzhou, Jiangsu
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Children's Hospital Of Fudan University, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No